# EFFECT OF EMDR 2.0 ONLÎNE GROUP PROTOCOL ON TRAUMATÎC EXPERÎENCES BASED ON TRAFFÎC ACCÎDENT: A RANDOMÎZED CONTROLLED TRÎAL

10/17/2022

### Study Protocol and Statistical Analysis Plan

To reach people who had been in car accidents, an announcement was posted on social media, the research was detailed, and volunteers were asked to give their contact information using Google Forms. The volunteers were interviewed and were thoroughly informed about the study, the inclusion requirements were assessed, and a Google Form information comprising data collecting tools will be delivered to the participants who fulfilled the inclusion criteria.

The subjects will be randomly divided into groups and the EMDR 2.0 Group application and mhGAP will be applied to them online. Participants eligible for the applications were randomized to be 30 subjects (in three group). In both groups, the application will bw made for three consecutive days. Those who will be unable to finish their applications at this stage will be ruled out of the study. Participants will be requested to complete out forms including data collection tools 1 week and 1 month after completing the applications. Following appropriate processing, the obtained data will be subjected to statistical analysis.

## **Statistical Analysis**

SPSS 22 package program will be used to perform statistical analyses on study data. Descriptive data will be presented with frequency and percentage for categorical variables and mean and standard deviation for continuous variables. The Pearson Chi-square test for categorical variables and parametric assumptions for continuous variables will be used to compare the pre-application variables of the two groups, followed by the Student's T-test. The repeated measures analysis of variance will be used to see whether EMDR 2.0 Group Application and mhGAP procedures alone resulted in significant changes in the dependent variables and if there will be a difference in changes between the two groups. In cases where the Mauchly test revealed that the sphericity assumption will be been violated, the Greenhouse–Geisser adjustment will be used, and the corrected results will be reported. The effect size will be determined using  $\eta 2$ . A value of p < 0.05 will be considered statistically significant.

#### **Data Collection Tools**

#### The Socio-Demographic Data Form

The socio-demographic data form will be developed by the researchers in line with the literature and study objectives. Participant's demographic data such as age, sex, educational level, and profession will be inquired.

#### The Depression-Anxiety-Stress Scale-21

The Depression-Anxiety-Stress Scale-21 (DASS-21) will be used in the study to determine the depression, anxiety, and stress symptoms of the participants. The scale has 21 items (Lovibond and Lovibond, 1995). Each question is evaluated on a four-point Likert-type scoring and it has seven items each for depression, anxiety, and stress. The score that can be obtained from the scale for each subdimension changes between 0 and 21. The Turkish validity and reliability study of the scale were conducted by Saricam (2018).

#### The Impact of Event Scale

The Impact of Event Scale (IES-R) will be applied to measure the amount of effect of persons from an event in the study. It was developed by Weis and Marmara in 1997 (Weiss, 2007). It is a self-report five-point Likert-type scale and includes 22 items. It evaluates the level of exposure to events in three different fields as "Intrusion," "Avoidance," and "Hyperarousal." The score that can be obtained from the scale varies between 0 and 88. The Turkish validity and reliability studies of the scale were carried out (Çorapçıoğlu et al., 2006).

#### **Informed Consent**

The purpose of this study is to decrease traumatic, depressive, and stressful symptoms of the people who experienced traffic accident through EMDR 2.0. It will be approximately 30 minutes to complete necessary questionnaires. The involvement of study is voluntarily basis, and you can be dismissed in any time of the study without losing any right.

After you sign this form, there will be relevant questions. The purpose of these questions to make comparison by a blind researcher in 1-week and 1-month follow up. All of the documents and information will be kept private, and there will be no publishing of this private information to the public. In case of publishing of the study findings, your identity will be kept private.

I read all of the information in the informed consent and accept to involve.



Figure 1. Flowchart of the study